CLINICAL TRIAL: NCT01344369
Title: A Study to Evaluate the Relative Bioavailability of Norethindrone/Ethinyl Estradiol 0.4 mg/0.035 mg Chewable Tablets (Teva Pharmaceuticals, USA) Compared to FEMCON® Fe (Norethindrone/Ethinyl Estradiol) 0.4 mg/0.035 mg Chewable Tablets (Warner Chilcott) in Healthy Female Volunteers Under Non-Fasted Conditions
Brief Title: Norethindrone/Ethinyl Estradiol 0.4 mg/35 Mcg Chewable Tablets Under Non-Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals, USA
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10816221
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Results first posted 2011-05-30 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Healthy Subjects; Bioequivalence
MeSH Terms: interventions — ovcon 35; Norethindrone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): Norethindrone/Ethinyl Estradiol 0.4 mg/0.035 mg Chewable Tablets (Teva)
  Interventions: Drug: Norethindrone/Ethinyl Estradiol
- Reference Listed Drug (Active Comparator): FEMCON® Fe 0.4 mg/0.035 mg Chewable tablets (Warner Chilcott)
  Interventions: Drug: FEMCON® Fe

INTERVENTIONS:
Drug: Norethindrone/Ethinyl Estradiol — 0.4 mg/0.035 mg Chewable Tablets
  Other Names: Zeosa®
  Arms: Investigational Test Product
Drug: FEMCON® Fe — 0.4 mg/0.035 mg Chewable Tablets
  Other Names: Ovcon® 35 Fe; norethindrone/ethinyl estradiol (generic name)
  Arms: Reference Listed Drug

SUMMARY:
The purpose of this study was to evaluate the relative bioavailability of a test formulation of norethindrone/ethinyl estradiol 0.4 mg/0.035 mg chewable tablets (Teva Pharmaceuticals, USA) compared to the reference listed product, FEMCON® Fe (norethindrone/ethinyl estradiol and ferrous fumarate) 0.4 mg/0.035 mg Chewable tablets (Warner Chilcott) under fed conditions in healthy, non-tobacco using, adult female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18-45 years of age inclusive with Body Mass Index within 18-30 kg/m2 inclusive, as described in Novum Standard Operating Procedures. Female subjects must either abstain from sexual intercourse or use a reliable non-hormonal method of contraception (e.g. condom with spermicide, diaphragm, non-hormonal IUD) from at least 14 days prior to the first study dosing, throughout the study, and until 14 days after the last dose.
* Normal menstrual cycle.
* Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
* Signed and dated informed consent form, which meets all criteria of current FDA regulations.

Exclusion Criteria:

* Post menopausal or have irregular menstrual cycle.
* Pregnant, lactating, or likely to become pregnant during the study.
* History of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* Significant history or current evidence of chronic infectious disease, system disorder, or organ dysfunction.
* Presence of gastrointestinal disease or history of malabsorption within the last year.
* History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
* Presence of a medical condition requiring regular treatment with prescription drugs.
* Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing.
* Participation in any clinical trial within 30 days prior to dosing.
* Drug or alcohol addiction requiring treatment in the past 12 months.
* Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days prior to dosing.
* Positive test results for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
* Positive test results for drugs of abuse at screening.
* Positive serum pregnancy test.
* Subjects who have ever had progestational hormone implants.
* Subjects who have had progestational hormone depot injections within 12 months proceeding dosing.
* Subjects who are using or have used within the 3 months preceding dosing any vaginally administered estrogen or progestin-containing products.
* Any personal or strong family history of estrogen- or progestogen-dependent tumors.
* History of clinically significant fibrocystic breast disease.
* Subjects with a history of thromboembolic disorders, myocardial infarction, or stroke.
* Use of norethindrone or ethinyl estrodiol-containing oral contraceptives within 30 days of initial dosing.
* Hysterectomy or oophorectomy (unilateral or bilateral)
* User of tobacco or nicotine containing products within 30 days of the start of the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Norethindrone/Ethinyl Estradiol (Test) First: 0.4 mg/0.035 mg Norethindrone/Ethinyl Estradiol 0.4 mg/0.035 mg Chewable Tablets test product dosed in first period followed by 0.4 mg/0.035 mg FEMCON® Fe Chewable Tablets reference product dosed in the second period.
- FEMCON® Fe (Reference) First: 0.4 mg/0.035 mg FEMCON® Fe Chewable tablets reference product dosed in first period followed by 0.4 mg/0.035 mg Norethindrone/Ethinyl Estradiol Chewable Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | FEMCON® Fe (Reference) First
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Washout of 28 Days
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | FEMCON® Fe (Reference) First
Started | 18 | 18
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Second Intervention
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | FEMCON® Fe (Reference) First
Started | 17 | 17
Completed | 17 | 16
Not Completed | 0 | 1
Not completed — Emesis within 2 x Tmax | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | FEMCON® Fe (Reference) First | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 12 | 14 | 26
  Caucasian | 2 | 1 | 3
  Hispanic | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Norethindrone
Description: Bioequivalence based on Norethindrone Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Norethindrone/Ethinyl Estradiol (Test): 0.4 mg/0.035 mg Norethindrone/Ethinyl Estradiol 0.4 mg/0.035 mg Chewable Tablets test product dosed in either period.
- FEMCON® Fe (Reference): 0.4 mg/0.035 mg FEMCON® Fe Chewable tablets reference product dosed in either period.
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | FEMCON® Fe (Reference)
Number analyzed (Participants) | 33 | 33
ng/mL | 4.3306 (1.7393) | 4.2282 (1.6696)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs FEMCON® Fe (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 102.44, 90% CI 2-sided [93.08 to 112.75] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Norethindrone
Description: Bioequivalence based on Norethindrone AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | FEMCON® Fe (Reference)
Number analyzed (Participants) | 33 | 33
ng*h/mL | 37.8065 (16.1921) | 37.3991 (15.3939)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs FEMCON® Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.58, 90% CI 2-sided [96.66 to 104.66] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Norethindrone
Description: Bioequivalence based on Norethindrone AUC0-inf (area under the concentration-time curve from time zero to infinity).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | FEMCON® Fe (Reference)
Number analyzed (Participants) | 33 | 33
ng*h/mL | 43.9982 (19.4559) | 43.8819 (18.8478)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs FEMCON® Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.85, 90% CI 2-sided [96.43 to 105.48] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax of Ethinyl Estradiol
Description: Bioequivalence based on Ethinyl Estradiol Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | FEMCON® Fe (Reference)
Number analyzed (Participants) | 33 | 33
pg/mL | 137.6758 (33.6231) | 137.8485 (37.6177)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs FEMCON® Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.59, 90% CI 2-sided [93.69 to 108.00] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: AUC0-t of Ethinyl Estradiol
Description: Bioequivalence based on Ethinyl Estradiol AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | FEMCON® Fe (Reference)
Number analyzed (Participants) | 33 | 33
pg*h/mL | 1916.2311 (433.4875) | 1987.6311 (478.7842)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs FEMCON® Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 96.68, 90% CI 2-sided [92.76 to 100.77] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: AUC0-inf of Ethinyl Estradiol
Description: Bioequivalence based on Ethinyl Estradiol AUC0-inf (area under the concentration-time curve from time zero to infinity).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | FEMCON® Fe (Reference)
Number analyzed (Participants) | 33 | 33
pg*h/mL | 2072.5423 (483.0176) | 2152.3775 (517.5977)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs FEMCON® Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 96.44, 90% CI 2-sided [92.22 to 100.84] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 6 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | FEMCON® Fe (Reference)
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 13/36 | 10/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norethindrone/Ethinyl Estradiol (Test) (N=36) | FEMCON® Fe (Reference) (N=36)
Abdominal Cramping (General disorders) | 4 (4) | 0 (0)
Sinus Congestion (General disorders) | 0 (0) | 2 (2)
Decreased Blood Pressure (General disorders) | 2 (2) | 2 (2)
Vomiting (General disorders) | 5 (5) | 3 (3)
Nausea (General disorders) | 6 (6) | 3 (3)
Headache (General disorders) | 5 (5) | 1 (1)
Increased Temperature (General disorders) | 0 (0) | 2 (2)
Increased Blood Pressure (General disorders) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.